CLINICAL TRIAL: NCT03119844
Title: Effects of Phototherapy Associated to Exercise-based Cardiac Rehabilitation Program in Chronic Heart Failure: Clinical Trial
Brief Title: Effects of Phototherapy Associated to Exercise-based Rehabilitation Program in Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Caroline Bublitz Barbosa, Principal Investigator, Federal University of São Paulo
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 54984116.6.0000.5505
Record Dates: First submitted 2017-04-11; First posted 2017-04-19 (Actual); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Heart Failure; Physical Activity
MeSH Terms: conditions — Heart Failure; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise and placebo phototherapy (Experimental): Placebo phototherapy and Cycle ergometer exercise rehabilitation protocol
  Interventions: Other: Exercise; Other: Placebo Phototherapy
- Exercise and active phototherapy (Experimental): Active phototherapy and Cycle ergometer exercise rehabilitation protocol
  Interventions: Other: Exercise; Other: Active Phototherapy

INTERVENTIONS:
Other: Exercise — The exercise will be performed in a cycle ergometer, intermittently, during 40 minutes, in a moderate intensity and prescribed by the perceived exertion Borg (PEB) scale.
Other: Placebo Phototherapy — Patients will receive the placebo application of low level laser therapy (parameters: 808nm, 100mW, 28J) in the rectus Femoris and gastrocnemius muscles of both lower limbs before the performance of the cycle ergometer exercise protocol.
  Arms: Exercise and placebo phototherapy
Other: Active Phototherapy — Patients will receive the active application of low level laser therapy (parameters: 808nm, 100mW, 28J) in the rectus Femoris and gastrocnemius muscles of both lower limbs before the performance of the cycle ergometer exercise protocol.
  Arms: Exercise and active phototherapy

SUMMARY:
Heart failure affects not only the cardiovascular system with structural abnormalities of the heart, but also the musculoskeletal system, leading to exercise intolerance. Objective: To evaluate the effects of a short-term exercise protocol and phototherapy, on the functional capacity and inflammatory markers in patients with heart failure. In addition, the investigators will investigate pulmonary function, peripheral and respiratory muscle strength and quality of life. Methods: Heart failure patients (left ventricular ejection fraction < 40%) will be selected from the outpatient clinic of the myocardium of the Department of Cardiology of Unifesp and randomized among two groups: patients who will be submitted to placebo phototherapy and cycle ergometer exercise; and patients who will be submitted to active phototherapy and cycle ergometer exercise. All groups will receive treatment twice a week for four weeks. Patients will be instructed to conduct home-based walking program at least twice a week. Patients will be evaluated before and after protocols regarding the pulmonary function, peripheral and respiratory muscle strength, functionality, quality of life and evaluation of systemic inflammatory mediators.

ELIGIBILITY:
Inclusion Criteria:

* Heart Failure diagnosis determined by clinical presentation and confirmed on echocardiography by clinicians, with a left ventricular ejection fraction (LVEF) < 40%
* New York Heart Association (NYHA) classes II and III.

Exclusion Criteria:

* chronic lung disease confirmed by pulmonary function testing
* unstable angina pectoris and acute coronary syndromes
* dialysis
* neuromuscular and psychiatric conditions that interfere in exercise

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Six-minute walk test to measure functional capacity change | Pre and post 4 weeks of rehabilitation programs
  According to the baseline distance walked, we will evaluate the improvement in functional capacity after the period of the rehabilitation programs
Inflammatory markers | Pre and post 4 weeks of rehabilitation programs
  Evaluate the change in levels of interleukin (IL): IL-1 and IL-10, and tumor necrosis factor-alpha (TNF-α)

SECONDARY OUTCOMES:
Respiratory muscle strength | Pre and post 4 weeks of rehabilitation programs
  By manovacuometry, assessing the change in inspiratory muscle pressure and expiratory muscle pressure
Peripheral muscle strength | Pre and post 4 weeks of rehabilitation programs
  By dynamometry, assessing the change in the peak force of quadriceps femoris muscle
Quality of life | Pre and post 4 weeks of rehabilitation programs
  By Minnesota Living with Heart Failure Questionnaire assessing the change in quality of life

OTHER OUTCOMES:
Six-minute walk test to measure functional capacity change | Follow up after 3 months of the end of the rehabilitation programs
  Evaluate the improvement in functional capacity
Respiratory muscle strength | Follow up after 3 months of the end of the rehabilitation programs
  By manovacuometry, assessing the change in inspiratory muscle pressure and expiratory muscle pressure
Peripheral muscle strength | Follow up after 3 months of the end of the rehabilitation programs
  By dynamometry, assessing the change in the peak force of quadriceps
Quality of life | Follow up after 3 months of the end of the rehabilitation programs
  By Minnesota Living with Heart Failure Questionnaire assessing the change in quality of life

IPD SHARING:
Plan to Share IPD: No